CLINICAL TRIAL: NCT00243373
Title: Using Barcode Technology to Improve Medication Safety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tejal Gandhi, Associate Professor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS14053-02
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Impact of Barcode Technology on Medication Errors
Keywords: Patient safety; Medication safety; Barcode technology

INTERVENTIONS:
Device: Barcode technology/eMAR

SUMMARY:
This study will investigate the impact of barcode technology on medication errors made by nursing. In addition, it will measure the impact of this technology on nursing workflow and satisfaction.

DETAILED DESCRIPTION:
Patient safety is a critical issue in healthcare1. Medications are the most commonly used form of medical therapy and the single most frequent cause of adverse events2. The medication use process has several stages: ordering, transcribing, dispensing, administering and monitoring. Medication errors have been shown to be common3,4, and a large proportion (61%) of them occur in the dispensing, transcribing and administering stages5. Barcode technology in conjunction with an electronic medication administration record (eMAR) system has been proposed as a promising way to reduce medication errors at the transcribing, dispensing, and administering stages6. However, its efficacy for reducing medication error rates, its acceptance by staff, and its cost-benefit ratio remain unknown. Without evidence to clarify these issues, it is difficult for health care organizations to prioritize this technology among many other potential safety interventions7. We therefore propose to answer 3 related questions in this study: i) What is the impact of barcode and electronic medication administration record (barcode/eMAR) technology on reducing medication errors in hospitalized patients? ii) What is the impact of barcode/eMAR technology on nursing and pharmacy efficiency and satisfaction? iii) Can the cost of barcode/eMAR technology be justified by its benefits? We propose to address these questions at the Brigham and Women's Hospital (BWH), which has a long-standing tradition of innovation in healthcare and research in medication safety. In particular, it was one of the first hospitals to assess the impact of computerized physician order entry (CPOE) on medication safety8,9. While CPOE is important for improving medication safety, it addresses errors primarily in the ordering stage of the medication use process, leaving patients vulnerable to errors that occur at the dispensing, transcribing and administering stages. Therefore, as part of a multi-disciplinary patient safety initiative, BWH has committed 3 million dollars to build a state-of-the-art barcode/eMAR system. This system will include sophisticated decision support to reduce medication errors made beyond the physician ordering stage. Design work is near completion and the hospital plans to implement the system in phases over 9 months beginning in the 4th quarter of 2003. This offers us a window of opportunity to formally study the broad impact of barcode/eMAR technology. We propose to perform a prospective, controlled, multidisciplinary randomized controlled trial of barcode/eMAR's impact on medication errors, as well as evaluations of impact on hospital efficiency, staff satisfaction, and hospital finances.

Specific Aims:

We plan to address the following 3 specific aims over the proposed 24 months of the study:

1. To evaluate the impact of barcode/eMAR technology on the rate of serious medication transcribing and administration errors.
2. To evaluate the impact of barcode/eMAR technology on nursing workflow and satisfaction in an acute care hospital.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who agree to be observed during the medication administration process before barcode technology
* Nurses who agree to be observed during the medication administration process after barcode technology is implemented

The goal is 6700 medication administration observations in the pre and the post periods

Exclusion Criteria:

* Nurses who refuse to be observed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6700 (Estimated)
Dates: Start 2005-04; Primary Completion 2005-12 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Transcription errors
Administration errors
Serious medication errors

SECONDARY OUTCOMES:
Nursing satisfaction
% nursing time spent on medication administration
ADEs

CONTACTS AND LOCATIONS:
Overall Officials: Tejal Gandhi, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Poon EG, Keohane CA, Yoon CS, Ditmore M, Bane A, Levtzion-Korach O, Moniz T, Rothschild JM, Kachalia AB, Hayes J, Churchill WW, Lipsitz S, Whittemore AD, Bates DW, Gandhi TK. Effect of bar-code technology on the safety of medication administration. N Engl J Med. 2010 May 6;362(18):1698-707. doi: 10.1056/NEJMsa0907115. PMID 20445181